CLINICAL TRIAL: NCT02740062
Title: A Novel Non Invasive Brain EEG Based Evaluation and Treatment for Central Manifestation Characteristics of Neuropathic Pain
Brief Title: Non Invasive Brain Evaluation and Treatment for Neuropathic Pain
Acronym: NIBSNP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NIBS NeuroScience Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Reuth-01
Record Dates: First submitted 2016-03-27; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment (Active Comparator): Active tDCS treatment
  Interventions: Device: NIBS system for evaluation and non invasive current stimulation
- Sham treatment (Sham Comparator): Sham tDCS treatment
  Interventions: Device: NIBS system for evaluation and non invasive current stimulation

INTERVENTIONS:
Device: NIBS system for evaluation and non invasive current stimulation

SUMMARY:
This trial is designed to preliminary evaluate the efficacy and safety of NIBS system for evaluation and treatment of neuropathic pain. The NIBS system evaluates brain neuronal network activity and customizes a personalized treatment utilizing low current non invasive brain stimulation technology for neuropathic pain with central component. this is single meeting trial which includes brain activity evaluation and a single treatment and sham treatment. The goal of the study is to evaluate the central brain component of neuropathic pain subjects, and the effect of conventional tDCS treatment.

DETAILED DESCRIPTION:
Neuropathic pain is a pain which persists after nerve injury has healed and results from significant functional and structural changes in the nervous system similar to memory processes. As a result, neuropathic pain has been proposed to be "a persistence of the memory of pain and/or the inability to extinguish the memory of pain evoked by an initial inciting injury". A firm conclusion in the neurobiology of learning and memory is that different types of memory have distinct mechanisms (e.g., declarative memory vs procedural memory). A similar distinction can be made in pain: various chronic pain states have distinct central mechanisms . Accumulating evidence suggests that chronic pain is a type of nociceptive memory mediated by structural and functional plasticity in by multiple pathways at cortical, subcortical, spinal, and peripheral levels.Elucidating the basal neuronal signature of the person suffering from chronic pain enables to optimizing a treatment which in all studies was constant for all patients regardless of their basal activity

In this study participants will undergo diagnosis of the personalized central manifestation characteristics of the neuropathic pain and evaluate the efficacy of a standard, most commonly used tDCS treatment, based on the diagnosis.

for this purpose a single meeting will take place during which participants will undergo evaluation, sham treatment and standard tDCS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic pain diagnosis by pain physician Up to 3 months before trial onset.
* Current NPRS>4

Exclusion Criteria:

* Neurological illness causing structural brain damage (e.g. Stroke, TIA)
* Psychiatric disease
* History of loss of consciousness
* Epilepsy or epilepsy in a first degree relative
* Medical implants
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain as measured by VAS (visual analog scale) | Before and 10 minutes after one time treatment
  VAS estimation before Treatment and 10 minutes after tDCS treatment.

SECONDARY OUTCOMES:
Von Frey sensitivity evaluation in neuropathic area | Before and 10 minutes after one time treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Reuth Medical Center, Tel Aviv, Other, Israel

IPD SHARING:
Plan to Share IPD: Undecided